CLINICAL TRIAL: NCT04411550
Title: A (Randomised, Double-Blind, Intravenous Single-Dose, Parallel, Four-Arm) Phase I Clinical Study to Compare Pharmacokinetics, Safety, and Immunogenicity of HLX11 vs. Perjeta® (US, EU, and CN-Sourced) in Healthy Chinese Male Subjects
Brief Title: Compare Pharmacokinetics, Safety, and Immunogenicity of HLX11 vs. Perjeta in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX11-001
Record Dates: First submitted 2020-05-19; First posted 2020-06-02 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HLX11 group (Experimental): HLX11 are given intravenous infusion at a single dose of 420 mg, and the administration time is 60 min (± 10 min).
  Interventions: Drug: HLX11
- CN-Perjeta group (Active Comparator): CN-Perjeta are given intravenous infusion at a single dose of 420 mg, and the administration time is 60 min (± 10 min).
  Interventions: Drug: CN-Perjeta(Pertuzumab)
- EU-Perjeta group (Active Comparator): EU-Perjeta are given intravenous infusion at a single dose of 420 mg, and the administration time is 60 min (± 10 min).
  Interventions: Drug: EU-Perjeta(Pertuzumab)
- US-Perjeta group (Active Comparator): US-Perjeta are given intravenous infusion at a single dose of 420 mg, and the administration time is 60 min (± 10 min).
  Interventions: Drug: US-Perjeta(Pertuzumab)

INTERVENTIONS:
Drug: HLX11 — healthy volunteers receive HLX11 (420mg) once
  Arms: HLX11 group
Drug: CN-Perjeta(Pertuzumab) — healthy volunteers receive CN-Perjeta (420mg) once
  Arms: CN-Perjeta group
Drug: EU-Perjeta(Pertuzumab) — healthy volunteers receive EU-Perjeta (420mg) once
  Arms: EU-Perjeta group
Drug: US-Perjeta(Pertuzumab) — healthy volunteers receive US-Perjeta (420mg) once
  Arms: US-Perjeta group

SUMMARY:
This is a randomised, double-blind, intravenous single-dose, four-arm parallel study designed to compare the PK of HLX11 and US, EU, and CN-sourced Perjeta® in healthy Chinese adult male subjects, and to assess the safety, tolerability, and immunogenicity of these 4 drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese males
* aged ≥ 18 and ≤ 45
* body mass index (BMI) ≥ 19 and ≤ 26 kg/m2
* LVEF≥ 55%

Exclusion Criteria:

* A history of any serious clinical disease such as haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, mental, neurological diseases, and tumour, or allergic diseases
* Use of a monoclonal antibody or any biological product within 6 months before study drug administration
* A history of allergic reactions or anaphylaxis, including such reactions to any drug or excipient in the clinical study
* Use of prescription drugs, over-the-counter drugs (OTC), or traditional Chinese medicine (TCM) (excluding vitamins, mineral supplements, and dietary supplements) within 28 days before study drug administration
* A history of blood donation within 3 months before study drug administration
* Participation in other clinical study and use of the investigational product/comparator within 3 months before study drug administration
* Positive for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody
* A history of drug abuse
* Failure to comply with protocol requirements, instructions, and study limitations, such as uncooperative attitude, failure to return to the study site for follow-up visits, or failure to complete the entire clinical study, as judged by investigators

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Cmax | from predose to 2352 hours (Day 99),13 timepoints
  Peak concentration
AUC0~t | from predose to 2352 hours (Day 99),13 timepoints
  Area under the plasma concentration-time curve from time 0 to the last concentration-measurable time point
AUC0~inf | from predose to 2352 hours (Day 99),13 timepoints
  Area under the plasma concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
safety and tolerability of 4 groups | from day1 to day 99
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
safety and tolerability of 4 groups | from day1 to day 99
  Number of AE as assessed by CTCAE v5.0
safety and tolerability of two groups | from day1 to day 99
  AE listing as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Principal Investigator — The Second Hospital of Anhui Medical University; Hui Zhao, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] American Society for Clinical Pharmacology and Therapeutics. Clin Pharmacol Ther. 2022 Mar;111 Suppl 1:S5-S80. doi: 10.1002/cpt.2521. No abstract available. PMID 35132630
- [Derived] Yang J, Lin L, Long Q, Zhang Q, Sun G, Zhou L, Wang Q, Zhu J, Li F, Hu W. HLX11, a Proposed Pertuzumab Biosimilar: Pharmacokinetics, Immunogenicity, and Safety Profiles Compared to Three Reference Biologic Products (US-, EU-, and CN-Approved Pertuzumab) Administered to Healthy Male Subjects. BioDrugs. 2022 May;36(3):393-409. doi: 10.1007/s40259-022-00534-w. Epub 2022 May 20. PMID 35594017